CLINICAL TRIAL: NCT00180453
Title: SPIRIT First: A Clinical Evaluation of an Investigational Device. The Abbott XIENCE V® Everolimus Eluting Coronary Stent System in the Treatment of Patients With de Novo Native Coronary Artery Lesions
Brief Title: SPIRIT FIRST Clinical Trial of the Abbott Vascular XIENCE V® Everolimus Eluting Coronary Stent System
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Matt Kiely, Abbott Vascular
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 02-350
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2010-01-06 (Estimated); Status verified 2009-06

CONDITIONS: Coronary Artery Disease; Everolimus; Vascular Disease; Myocardial Ischemia; Coronary Artery Stenosis
Keywords: Cardiovascular disease; Ischemia
MeSH Terms: conditions — Coronary Artery Disease; Vascular Diseases; Myocardial Ischemia; Coronary Stenosis; Cardiovascular Diseases; Ischemia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Abbott Vascular XIENCE V® Everolimus Eluting Coronary Stent System
  Interventions: Device: Coronary artery drug eluting stent placement
- 2 (Active Comparator): Abbott Vascular MULTI-LINK VISION® BMS
  Interventions: Device: Coronary artery stent placement

INTERVENTIONS:
Device: Coronary artery drug eluting stent placement — Coronary artery drug eluting stent placement
  Arms: 1
Device: Coronary artery stent placement — Coronary artery stent placement
  Other Names: Abbott Vascular MULTI-LINK VISION® coronary stent system
  Arms: 2

SUMMARY:
Prospective, randomized, controlled, single-blinded, parallel two-arm, multicenter trial.

Test arm: XIENCE V® Everolimus Eluting Coronary Stent System(stent length: 18mm, diameter: 3.0mm) Control arm: Metallic stent (MULTI-LINK VISION® metallic stent(stent length: 18mm, diameter: 3.0mm) Follow-up angiographic imaging and intra vascular ultra sound (IVUS) at 180 days and 1 year

DETAILED DESCRIPTION:
The SPIRIT FIRST clinical trial will enroll approximately 60 patients and will assess the feasibility and performance of the XIENCE V® Everolimus Eluting Coronary Stent System in the treatment of patients with de novo native coronary artery lesions. In this trial, the XIENCE V® Everolimus Eluting Coronary Stent System will be compared to the MULTI-LINK VISION® metallic stent which is CE marked and FDA approved and is available for commercial use in Europe and in the United States. The SPIRIT FIRST Clinical trial will enroll approximately 60 patients (30 patients in the test arm and 30 patients in the control arm) with de novo native coronary artery lesions in 4 clinical sites in The Netherlands and Germany

ELIGIBILITY:
Inclusion Criteria

1. Patient must be at least 18 years of age.
2. Patient is able to verbally acknowledge an understanding of the associated risks, benefits and treatment alternatives of receiving the XIENCE™ V Everolimus Eluting Coronary Stent System and his or her legally authorized representative provides written informed consent prior to the stent procedure, as approved by the appropriate Ethics Committee.
3. Patient must have evidence of myocardial ischemia (e.g., stable or unstable angina, silent ischemia, positive functional study).
4. Patient must be an acceptable candidate for coronary artery bypass graft (CABG) surgery.
5. Patient must agree to undergo all protocol-required follow-up examinations including angiographic and IVUS follow-up at two time points (180 days and 1 year ).
6. Female patients of childbearing potential must have had a negative pregnancy test within 7 days before treatment, and must not be nursing at the time of treatment.
7. Female patients of childbearing potential must also agree at time of consent to use birth control up to and including the second angiographic follow-up at 1 year.

Inclusion Criteria: Angiographic

1. Planned single, de novo, type A - B1, native coronary artery lesion treatment.
2. Target lesion must be located in a native vessel with a diameter of 3.0 mm assessed by QCA on-line.
3. Target lesion length ≤ 12 mm, assessed by QCA on-line.
4. The target lesion must be in a major artery or branch with a stenosis of ≥ 50% and < 100% assessed by QCA on-line and with a TIMI flow of ≥ 1.

Exclusion Criteria

1. Patient has had a known acute myocardial infarction (greater than two times the upper limit of normal CK with presence of CK-MB) within 3 days preceding the index procedure and CK has not returned to normal limits at the time of the procedure.
2. Patient has current or a history of unstable arrhythmias, regardless of whether cardiac rhythm management devices are used (e.g., pacemaker, Automatic Implantable Cardioverter Defibrillator).
3. Patient has a known left ventricular ejection fraction ≥ 30%.
4. Patient has received a heart transplant or any other organ transplant or is on a waiting list for any organ transplant.
5. Patient is receiving or scheduled to receive chemotherapy or radiation therapy within 30 days prior to or after the procedure.
6. Patient is receiving immunosuppression therapy or has known immunosuppressive disease.
7. Patient is receiving chronic anticoagulation therapy (e.g., heparin, coumadin).
8. Patient has a known hypersensitivity or contraindication to aspirin, heparin, clopidogrel, cobalt, chromium, nickel, tungsten, everolimus, acrylic and fluoro polymers or contrast sensitivity that cannot be adequately pre-medicated.
9. Patient has a platelet count <100,000 cells/mm3 or >700,000 cells/mm3, a WBC of <3,000 cells/mm3, or documented or suspected liver disease (including laboratory evidence of hepatitis).
10. Patient has known renal insufficiency (e.g., serum creatinine level of more than 2.5 mg/dL, patient on dialysis).
11. Patient has a history of bleeding diathesis or coagulopathy or will refuse blood transfusions.
12. Patient has had a cerebrovascular accident (CVA) or stroke or transient ischemic neurological attack (TIA) within the past six months.
13. Patient has had a significant GI or urinary bleed within the past six months.
14. Patient has extensive peripheral vascular disease that precludes safe 6 French sheath insertion or extreme anticoagulation.
15. Patient has other medical illness (e.g., cancer or congestive heart failure) or recent history of substance abuse that may cause non-compliance with the protocol, confound the data interpretation or is associated with a limited life expectancy (i.e., less than one year).
16. Patient is already participating in another investigational use device or drug study or has completed the follow-up phase of another trial within the last 30 days.
17. Patient has received a drug eluting stent within the last 1 year.

Exclusion Criteria: Angiographic

1. The target lesion meets any of the following criteria:

   1. Aorto-ostial location
   2. Unprotected left main location
   3. Located within 2 mm of the origin of the LAD or LCX
   4. Located within or distal to an arterial or saphenous vein graft
   5. Located within 2 mm of a bifurcation
   6. Located distal to a previously implanted stent (same major epicardial vessel)
   7. Located in a major epicardial vessel that has been previously treated with brachytherapy
   8. Located in a major epicardial vessel that has been previously treated with any type of PCI (e.g., POBA, stent, cutting balloon, atherectomy), except if previous treatment occurred in a side branch distal to target lesion at least 180 days preceding the index procedure
   9. Involves jailing of side branches > 2.0 mm in diameter
   10. Total occlusion (TIMI flow 0)
   11. Excessive tortuosity proximal to or within the lesion
   12. Extreme angulation (≥ 90%) proximal to or within the lesion
   13. Moderate to heavy calcification
   14. Restenotic from previous intervention
2. The target vessel contains thrombus.
3. Another significant lesion (≥ 40 %DS) is located in the same major epicardial vessel as the target lesion.
4. Patient has a high probability that a procedure other than pre-dilatation and stenting will be required for treatment of the target vessel (e.g. atherectomy, cutting balloon).
5. Patient has additional lesion(s) for which an intervention within 180 days (prior to or after) of the index procedure would be required or has been performed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2003-12; Primary Completion 2005-04 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
In-stent late loss | at 180 days post procedure

SECONDARY OUTCOMES:
In-stent late loss | at 1 year post procedure
In-segment Late Loss | at 180 days and 1 year
In-stent and in-segment %Volume Obstruction | at 180 days and 1 year
In-stent and in-segment %Diameter Stenosis | at 180 days and 1 year
In-stent and in-segment Angiographic Binary Restenosis rate | at 180 days and 1 year
Persisting incomplete apposition, late incomplete apposition, aneurysm, thrombus, persisting dissection | at 180 days and 1 year
Major Adverse Cardiac Events | at 30, 180, 270 days, and 1, 2, 3, 4, 5 years
Target Vessel Failure | at 30, 180, 270 days, and 1, 2, 3, 4, 5 years
Acute success (device, procedure and clinical) | Acute

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Serruys, MD, Principal Investigator — Erasmus Medical Center
Locations (7):
- Skejby Sygehus, Aarhus, Denmark
- Germany (4):
  - Herzzentrum Bad Krozingen, Bad Krozingen
  - Kerckhoff-Klinik, Bad Nauheim
  - Herzzentrum Bad Oeynhausen, Bad Oeynhausen
  - Herzzentrum Siegburg GmbH, Siegburg
- Netherlands (2):
  - Academisch Medisch Centrum, Amsterdam
  - Erasmus Medical Center, Rotterdam

REFERENCES:
- [Background] Tsuchida K, Garcia-Garcia HM, Ong AT, Valgimigli M, Aoki J, Rademaker TA, Morel MA, van Es GA, Bruining N, Serruys PW. Revisiting late loss and neointimal volumetric measurements in a drug-eluting stent trial: analysis from the SPIRIT FIRST trial. Catheter Cardiovasc Interv. 2006 Feb;67(2):188-97. doi: 10.1002/ccd.20581. PMID 16400664
- [Result] Popma JJ, Tulli M. Spirit First - Another hurdle is cleared. EuroIntervention. 2005 Nov;1(3):260-3. No abstract available. PMID 19758913
- [Result] Serruys PW, Ong AT, Piek JJ, Neumann FJ, van der Giessen WJ, Wiemer M, Zeiher A, Grube E, Haase J, Thuesen L, Hamm C, Otto-Terlouw PC. A randomized comparison of a durable polymer Everolimus-eluting stent with a bare metal coronary stent: The SPIRIT first trial. EuroIntervention. 2005 May;1(1):58-65. PMID 19758878
- [Result] Tsuchida K, Piek JJ, Neumann FJ, van der Giessen WJ, Wiemer M, Zeiher AM, Grube E, Haase J, Thuesen L, Hamm CW, Veldhof S, Dorange C, Serruys PW. One-year results of a durable polymer everolimus-eluting stent in de novo coronary narrowings (The SPIRIT FIRST Trial). EuroIntervention. 2005 Nov;1(3):266-72. PMID 19758915
- [Result] SPRITI FIRST: 2-Jahres-ergebnisse. A durable polymer everolimus-eluting stent in de novo coronary narrowings. Richartz B.; Silber S. Herz ( Germany ) June 1, 2006 , 31/4 (359). ISSN: 0340-9937. Language: German
- [Derived] Muramatsu T, Onuma Y, van Geuns RJ, Chevalier B, Patel TM, Seth A, Diletti R, Garcia-Garcia HM, Dorange CC, Veldhof S, Cheong WF, Ozaki Y, Whitbourn R, Bartorelli A, Stone GW, Abizaid A, Serruys PW; ABSORB Cohort B Investigators; ABSORB EXTEND Investigators; SPIRIT FIRST Investigators; SPIRIT II Investigators; SPIRIT III Investigators; SPIRIT IV Investigators. 1-year clinical outcomes of diabetic patients treated with everolimus-eluting bioresorbable vascular scaffolds: a pooled analysis of the ABSORB and the SPIRIT trials. JACC Cardiovasc Interv. 2014 May;7(5):482-93. doi: 10.1016/j.jcin.2014.01.155. Epub 2014 Apr 16. PMID 24746650